CLINICAL TRIAL: NCT06062212
Title: Effect of Transpulmonary Mechanical Power on the Prognosis of Patients With Severe Acute Respiratory Distress Syndrome Treated With Venovenous Extracorporeal Membrane Oxygenation
Brief Title: Effect of Transpulmonary MP on Prognosis of Patients With Severe ARDS Treated With VV-ECMO
Status: Recruiting | Type: Observational
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Rui Wang, Principal Investigator, Beijing Chao Yang Hospital
Other Study IDs: 2023-KE-926
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Acute Respiratory Distress Syndrome; Extracorporeal Membrane Oxygenation; Mechanical Power; Transpulmonary Mechanical Power
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Arterial blood gas analysis, blood routine, liver and kidney function, coagulation, and BNP
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Transpulmonary pressure group
  Interventions: Procedure: Transpulmonary pressure

INTERVENTIONS:
Procedure: Transpulmonary pressure — Use transpulmonary pressure to guide ventilator setting in ECMO for severe ARDS patients.

SUMMARY:
Venovenous extracorporeal membrane oxygenation (VV-ECMO) is a salvage treatment for severe acute respiratory distress syndrome (ARDS). With the large-scale implementation of VV-ECMO in critical care medicine departments in China, significant progress has been made in treating severe ARDS. However, the patient mortality rate remains high. The pathophysiological essence of ARDS is an imbalance between the body's oxygen supply and demand, causing tissue and cell hypoxia, organ dysfunction, and even death. The VV-ECMO treatment process still requires mechanical ventilation assistance. However, inappropriate mechanical ventilation settings can lead to ventilator-related lung injury (VILI). In recent years, mechanical power has gradually attracted everyone's attention and is considered the cause of VILI. The transpulmonary mechanical power is more accurate to the energy directly performed to the lung tissue. Transpulmonary mechanical energy has a specific value in judging the prognosis of mechanically ventilated patients, but its clinical significance in treating patients with VV-ECMO is unclear. This study aimed to explore the value of transpulmonary mechanical power in predicting the prognosis of patients with severe ARDS patients treated with VV-ECMO.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of Berlin's definition for ARDS;
2. Receiving VV-ECMO support.

Exclusion Criteria:

1. Patients had been on high pressure (Ppeak >35 cm H2O) and a high fraction of inspired oxygen (FiO2>0.8) ventilation for >7 days;
2. Patients had a contraindication to heparinization;
3. Patients had an irreversible neurological injury;
4. Patients had severe chronic lung disease with life expectancy <6 months.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Severe ARDS patients treated with VV-ECMO
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patients successfully weaned from VV-ECMO | After patients enrolled 60 days
  Weaning VV-ECMO more than 48 hours with stable oxygenation and no need to re-establish ECMO

SECONDARY OUTCOMES:
60-day mortality | After patients enrolled 60 days
  Mortality rate at 60 days of VV-ECMO support

CONTACTS AND LOCATIONS:
Overall Officials: Rui Wang, Dr., Study Director — Beijing Chao-Yang Hospital, Capital Medical University, Beijing, China
Locations (1):
- Beijing Chao-Yang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No